CLINICAL TRIAL: NCT02579746
Title: Dietary Approach to Stop Hypertension With Sodium (Na) Reduction for Chinese Canadians
Acronym: DASHNa-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Ping Zou, RN PhD, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UofT30496
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: hypertension; immigrant; dietary intervention; lifestyle modification
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): The intervention group received usual care plus the DASHNa-CC intervention.
  Interventions: Behavioral: DASHNa-CC; Behavioral: usual care
- control (Active Comparator): The control group received usual care.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: DASHNa-CC — The 8-week DASHNa-CC intervention incorporated Dietary Approach to Stop Hypertension (DASH) diet, sodium reduction with the food therapy of Traditional Chinese Medicine, and included an intervention manual, two sessions of classroom instruction delivered in Mandarin, and a 20-minute telephone follow-up.
  Arms: intervention
Behavioral: usual care — education booklet, encouragement of physician visit, use of public health resources if needed

SUMMARY:
The study examined the feasibility of the Dietary Approach to Stop Hypertension with Sodium (Na) Reduction for Chinese Canadian (DASHNa-CC) intervention and its potential effects on blood pressure, health-related quality of life, and health service utilization. Half of participants received usual care while the other half received the DASHNa-CC intervention.

DETAILED DESCRIPTION:
Hypertension has been identified as the most important risk factor for cardiovascular diseases and accounts for a large proportion of stroke, myocardial infarction and heart failure in the Chinese population. While unhealthy diet has been identified as a modifiable risk factor for hypertension, there is a lack of culturally sensitive dietary intervention targeting Chinese Canadians. The 8-week DASHNa-CC intervention incorporated Dietary Approach to Stop Hypertension (DASH) diet, sodium reduction with the food therapy of Traditional Chinese Medicine, and included an intervention manual, two sessions of classroom instruction delivered in Mandarin, and a 20-minute telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* were at least 45 years old;
* had a systolic blood pressure 140 to 159 mmHg, or a diastolic blood pressure 90 to 99 mmHg, based on pre-intervention baseline assessment;
* were able to understand (listen) and speak in Mandarin, read and write in Chinese; and
* had access to a telephone.

Exclusion Criteria:

* used antihypertensive medications or other medications that raise or lower blood pressure during the previous three months;
* used TCM or professional TCM counselling to decrease blood pressure during the previous three months;
* used insulin or oral hypoglycemic agents during the previous three months;
* had a history of a cardiovascular event (stroke, myocardial infarction, percutaneous transluminal coronary angioplasty, coronary artery bypass surgery, or other arteriosclerotic cardiovascular disease related therapeutic procedure) during the previous three months;
* had a history of congestive heart failure;
* had a cancer diagnosis or treatment during the past two years;
* had special dietary requirements;
* were pregnant, breast feeding, or planned for pregnancy prior to the anticipated end of study;
* were a household member of another DASHNa-CC participant; or
* planned to leave the area prior to the anticipated end of study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
blood pressure | 8 weeks post randomization
  systolic and diastolic blood pressure

SECONDARY OUTCOMES:
health related quality of life | 8 weeks post randomization
  used SF-36v2